CLINICAL TRIAL: NCT00058955
Title: Physiological, Behavioral and Subjective Effects of Drugs (GHB)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orphan Medical (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Senior Director of Clinical Development, Jazz Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OMC-SXB-25; BPR00-09-27-02
Record Dates: First submitted 2003-04-15; First posted 2003-04-16 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Sedative Abuse
Keywords: ghb; Xyrem; triazolam; pentobarbital; sedative; abuse
MeSH Terms: interventions — Sodium Oxybate; Triazolam; Pentobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Sodium oxybate
  Interventions: Drug: sodium oxybate, triazolam and pentobarbital
- 2 (Active Comparator): triazolam
  Interventions: Drug: sodium oxybate, triazolam and pentobarbital
- 3 (Active Comparator): pentobarbital
  Interventions: Drug: sodium oxybate, triazolam and pentobarbital
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: sodium oxybate, triazolam and pentobarbital

INTERVENTIONS:
Drug: sodium oxybate, triazolam and pentobarbital — sodium oxybate, triazolam and pentobarbital
  Other Names: Xyrem

SUMMARY:
The purpose of this study is to learn more about the effects of gamma-hydroxybutyric acid (GHB) by comparing its physiological, behavioral and subjective effects with those of several other drugs.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about the effects of gamma-hydroxybutyric acid by comparing its physiological, behavioral and subjective effects with those of several other drugs.

This trial will be conducted as a double-blind, double-dummy, placebo-controlled, counter-balanced (Latin-square design) crossover study in volunteers with histories of sedative abuse. Volunteers will be recruited through advertising and word-of-mouth.

Volunteers will reside on our residential research unit for the duration of the study and participate in a maximum of 16 experimental sessions. Sessions will be conducted five days a week (Monday through Friday). The primary subjective and behavioral measures will be taken before drug administration and at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after drug administration.

ELIGIBILITY:
INCLUSION CRITERIA

* are ages 18-50 years
* have histories of sedative (e.g., GHB, alcohol, benzodiazepine or barbiturate) abuse
* are within 20% of their ideal body weight
* are healthy as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, and routine medical blood and urinalysis laboratory tests
* are not currently pregnant or breast-feeding, if female
* have signed and dated an informed consent form prior to beginning the study
* are willing and able to participate

EXCLUSION CRITERIA

* have a history or current serious medical or psychiatric conditions, including (but not limited to): heart condition, lung disease, diabetes, seizure disorders, significant gastrointestinal disturbances, narrow angle glaucoma, ulcers, sleep apnea, schizophrenia, personality disorder, bipolar disorder, paranoia, multiple personality disorder
* have hypersensitivity/allergy or other contraindications to sedatives or stimulants
* are physically dependent on alcohol or other drugs, excluding nicotine and caffeine
* are females who are pregnant or are breast feeding
* are females who become pregnant during the study as evaluated using periodic pregnancy tests

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-08; Study Completion 2005-03

PRIMARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Roland Griffiths, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine/Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860